CLINICAL TRIAL: NCT06569082
Title: CD34+ Selected Donor Cell Boost for Management of Poor Graft Function or Primary or Secondary Graft Failure Following Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: CD34+ Selected Stem Cell for Poor Graft Function or Graft Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-00885
Record Dates: First submitted 2024-08-22; First posted 2024-08-23 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Graft Failure; Poor Graft Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Individuals with Poor Graft Function or Failure Following Allogeneic HSCT (Experimental): The recipient will undergo evaluations, then undergo a single infusion of CD34 selected HSCT from the original donor.
  No additional GvHD prophylaxis will be administered. Patients who develop GvHD will receive the standard of care based on the discretion of the treating physician .
  Patients will receive supportive care per institutional standards and at the discretion of the treating physician.
  Interventions: Device: CD34+ Selected Donor Cell Boost; Procedure: Blood Stem Cell Infusion

INTERVENTIONS:
Device: CD34+ Selected Donor Cell Boost — The CliniMACS CD34 Reagent System is used to separate CD34 cells from the remaining stem cell product, using a peripheral blood stem cell sample provided by the original donor. These CD34 cells are then infused into the recipient following selection with the intent to restore function of the blood forming cells.
  Other Names: CliniMACS CD34 Reagent System
Procedure: Blood Stem Cell Infusion — The selected CD34 cells separated by the CliniMACS CD34 Reagent System are infused into the recipient.

SUMMARY:
The proposed trial is a single arm, non-randomized, single center pilot study utilizing CliniMACS CD34 Reagent System for patients following allogeneic hematopoietic stem cell transplant (HSCT) requiring treatment of graft dysfunction or failure.

DETAILED DESCRIPTION:
The primary objective of the study is to estimate the incidence of engraftment with sustained recovery of blood counts, including, absolute neutrophil cell (ANC) and platelet engraftment.

* ANC engraftment is defined as ANC of ≥ 0.5 × 10^9/L for three consecutive laboratory values obtained on different days. Date of ANC recovery is the date of the first of three consecutive laboratory values where the ANC is ≥ 0.5 × 10^9/L.
* Platelet engraftment should reflect no platelet transfusions administered for seven consecutive days. Report the date of the first of three consecutive laboratory values ≥ 20 × 10^9/L obtained on different days.

The secondary objective of the study is to estimate the incidence of Graft-versus-host disease (GvHD) and side effects that can be attributed to the CliniMACS CD34 Selected Cellular Product.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of allogeneic transplantation, adult ≥18 years, from any type of donor including matched related, matched unrelated, mismatched related or mismatched unrelated or haploidentical donor transplant.
* Documented evidence of graft dysfunction or failure (a-c):

  1. Primary graft Failure: Graft failure is defined as failure to achieve neutrophil engraftment by day +28 or lack of donor chimerism > 50% by day 45 not due to the underlying malignancy;
  2. Poor graft function is defined by at least 2 of the following 3 criteria: Hemoglobin < 8 g/dL, ANC < 0.5x109/L, and platelets < 20x109/L. The cytopenia must be unexplained (such as by disease relapse) and unresponsive to hematopoietic growth factors and must last at least 4 weeks;
  3. Secondary graft failure is defined as poor graft function associated with donor chimerism < 5% after initial engraftment
* Transplanted donor availability
* Negative pregnancy test within seven (7) days of product infusion for women of childbearing potential.

Exclusion Criteria:

* Graft failure due to disease relapse or evidence of disease relapse or progression
* Donor unavailable or unable to collect peripheral HPC by apheresis
* Responsive to conventional measures (such as, hematopoietic growth factor)
* Allergic reaction to murine proteins or iron dextran
* Women of childbearing potential with positive serum HCG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2034-08 (Estimated); Study Completion 2035-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Absolute Neutrophil Cell (ANC) Engraftment | Day 100 Post-Procedure
  ANC engraftment is defined as ANC of ≥ 0.5 × 10^9/L for three consecutive laboratory values obtained on different days.
Number of Participants with Platelet Engraftment | Day 100 Post-Procedure
  Platelet engraftment is defined as no platelet transfusions administered for seven consecutive days.

SECONDARY OUTCOMES:
Number of Participants with Grade II-IV Acute GVHD | Day 100 Post-Procedure
  The diagnosis of acute GvHD is based on clinical and pathological evaluation by the principal investigator in collaboration with the treating physician.
Number of Participants with Moderate to Severe Chronic GVHD | Day 365 Post-Procedure
  The diagnosis of chronic GvHD is based on clinical and pathological evaluation by the principal investigator in collaboration with the treating physician.

CONTACTS AND LOCATIONS:
Overall Officials: Jingmei Hsu, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, will be shared upon reasonable request provided the investigator whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose executes a data use agreement with NYU Langone Health. Requests may be directed to: Jingmei.hsu@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: No time limit.
Access Criteria: Requests should be directed to Jingmei.hsu@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.